CLINICAL TRIAL: NCT04194437
Title: Prospective Trial to Evaluate the Effectiveness of The Portable Organ Care System (OCS) Liver for Preserving, Optimizing and Assessing Currently Seldom Utilized DCD Donor Livers for Transplantation
Brief Title: OCS Liver DCD Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment in Liver DCD was stopped as a result of the FDA approval for the OCS Liver System and follow-up ended on 12/16/2024 based on adequate patient follow-up.
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LVR-092019
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- OCS Preserved Livers (Experimental): This is a single-arm trial of OCS preserved livers used for transplantation.
  Interventions: Device: OCS Liver System

INTERVENTIONS:
Device: OCS Liver System — The OCS Liver System will be used to preserve, optimize and assess livers from DCD donors.

SUMMARY:
Evaluate the safety and effectiveness of the OCS Liver System to preserve, optimize the condition, and assess levers from DCD donors.

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of the OCS™ Liver to preserve, optimize the condition and assess livers from DCD donors that currently are seldom used for liver transplants due to limitations of cold static storage with extended warm ischemic time and older donors.

ELIGIBILITY:
Inclusion Criteria:

* Registered primary liver transplant candidate
* Age ≥ 18 years
* Obtained informed consent

Exclusion Criteria:

* Acute, fulminant liver failure
* Prior solid organ or bone marrow transplant
* Ventilator dependent on day of transplant/donor organ offer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elbetanony, MD, Study Director — TransMedics
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mount Sinai Hospital, New York, New York
  - University of Texas San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Kubal C, Mihaylov P, Holden J. Oncologic indications of liver transplantation and deceased donor liver allocation in the United States. Curr Opin Organ Transplant. 2021 Apr 1;26(2):168-175. doi: 10.1097/MOT.0000000000000866. PMID 33650998

RESULTS

PARTICIPANT FLOW:
Groups:
- OCS Preserved Livers: OCS Liver System: OCS Liver System for preserving and assessing donor livers for transplantation from DCD donors.
Period: Overall Study
Arm/Group | OCS Preserved Livers
Started | 9
Completed (Completing the 6 month visit.) | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OCS Preserved Livers
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Liver Graft Survival Through 6 Months Post-transplant
Description: Evaluation of graft survival as defined per UNOS data collection criteria for graft status after liver transplantation
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preserved Livers
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: Liver graft-related serious adverse events (LGRSAEs) were collected up to the 30-day follow-up after transplantation. Ischemic biliary cholangiopathy was collected at 6 months post-transplant. Reporting of all-cause mortality is through 6-months post transplant.
Description: Per the protocol only liver graft-related serious adverse events (LGRSAEs) and serious adverse events (SAEs) will be collected through Day 30 post-transplant. Ischemic biliary cholangiopathy was collected at 6 months post-transplant.
  Other (Not Including Serious) Adverse Events were not collected and therefore not reported.
Arm/Group | OCS Preserved Livers
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Preserved Livers (N=9)
Intra-abdominal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic Artery Dissection (Vascular disorders) | 1 (1)
Ischemic Biliary Stricture (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall have right to publish results. To balance this right with TransMedics' (TM proprietary interests, site will submit manuscripts intended for publication for TM's review at least 30d prior to submission date. TM will complete its review within 30d of receipt. TM may request that site delete from its manuscripts any reference to TM confidential information and site shall promptly comply with such request. After 60d period, site will have right to publish manuscript, as amended by TM.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT04194437/Prot_SAP_000.pdf